CLINICAL TRIAL: NCT00831909
Title: Epidemiological Study to Describe Non-small Cell Lung Cancer (NSCLC) Clinical Management Patterns in Europe. Lung
Brief Title: Epidemiological Study to Describe NSCLC Clinical Management Patterns in Europe. Lung-EPICLIN
Acronym: EPICLIN
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Nadia Badri, European Medical Affairs Director Oncology, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-OEU-DUM-2008/1
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: NSCLC
Keywords: Lung Cancer; NSCLC management; NSCLC use of health care resources
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All NSCLC patients attending the responsible department of treating this type of patients (e.g. Oncology Department, Pneumology Department) for the first time (regardless of whether the patient is diagnosed with locally, advanced or metastatic disease) at the participating sites from the first of January 2009 to the end of March 2009. Patients diagnosed, or even treated, in other departments within the same hospital or in another hospital are susceptible to be included in the study if full access to the patient's medical record is made available.

SUMMARY:
To provide accurate and reliable information regarding NSCLC clinical management across European countries in order to detect unmet medical needs of this disease in terms of: patient and hospital characteristics; diagnostic and treatment approaches: initial and subsequent, follow-up patterns in clinical management; outcomes: symptoms, death, functionality, quality of life; use of resources and burden on patients and health care systems.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed NSCLC diagnosis (e.g. bronchoscope or FNAB), all stages, men and women, attending the responsible department of treating this type of patients for the first time between January 1st, 2009 and March 31st, 2009.
* For PRO sub-sample: ability to read and write since they will be asked to participate in the PRO part of the study. Selection will not be based on the disease stage of each patient, in order to avoid a selection bias.

Exclusion Criteria:

* According to the study design there will not be any exclusion criteria in order to provide a high external validity and to obtain the most accurate real daily practice information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All NSCLC patients attending the responsible department of treating this type of patients (e.g. Oncology Department, Pneumology Department) for the first time (regardless of whether the patient is diagnosed with locally, advanced or metastatic disease) at the participating sites from the first of January 2009 to the end of March 2009. Patients diagnosed, or even treated, in other departments within the same hospital or in another hospital are susceptible to be included in the study if full access to the patient's medical record is made available.
Sampling Method: Probability Sample
Enrollment: 3513 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To provide accurate, reliable information on NSCLC clinical management across European countries in order to detect unmet medical needs of this disease | 1 year follow up

SECONDARY OUTCOMES:
To assess the differences in patient characteristics, disease stage (differentiating between non-advanced disease, locally advanced disease, metastatic disease), and in clinical management across European countries. | 1 year follow up
To detect differences in clinical outcomes and related factors among countries. | 1 year follow up
To identify factors associated with clinical outcomes (patient, disease stage and clinical management related factors): predictive modelling for improved patient outcome. | 1 year follow up
To identify factors associated with the different levels of functional status and quality of life. | 1 year follow up
To compare the use of health care resources among countries. | 1 year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Carrato, MD, Principal Investigator — Hospital Ramón y Cajal, Madrid (Spain); Esteban Medina, Study Director — Medical Department, AstraZeneca Spain
Locations (162):
- Belgium (5):
  - Research Site, Antwerp
  - Research Site, Brussels
  - Research Site, Genk
  - Research Site, Herstal
  - Research Site, Liège
- France (76):
  - Research Site, Aix-en-Provence
  - Research Site, Ambilly
  - Research Site, Antibes
  - Research Site, Aulnay-sous-Bois
  - Research Site, Bar-le-Duc
  - Research Site, Beauvais
  - Research Site, Beuvry
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Cahors
  - Research Site, Castelnau-le-Lez
  - Research Site, Chalon-sur-Saône
  - Research Site, Chauny
  - Research Site, Chevilly-Larue
  - Research Site, Cholet
  - Research Site, Clamart
  - Research Site, Colmar
  - Research Site, Compiègne
  - Research Site, Coulommiers
  - Research Site, Denain
  - Research Site, Dijon
  - Research Site, Douai
  - Research Site, Draguignan
  - Research Site, Épinal
  - Research Site, Flers
  - Research Site, Givors
  - Research Site, Granville
  - Research Site, Grasse
  - Research Site, Guingamp
  - Research Site, Hyères
  - Research Site, Jonzac
  - Research Site, La Ferté-Bernard
  - Research Site, La Rochelle
  - Research Site, La Tronche
  - Research Site, Le Mans
  - Research Site, Liévin
  - Research Site, Limoges
  - Research Site, Longjumeau
  - Research Site, Lyon
  - Research Site, Mantes-la-Jolie
  - Research Site, Martigues
  - Research Site, Meaux
  - Research Site, Metz
  - Research Site, Metz-Tessy
  - Research Site, Mont-de-Marsan
  - Research Site, Mont-Saint-Martin
  - Research Site, Montpellier
  - Research Site, Moulins
  - Research Site, Mulhouse
  - Research Site, Nancy
  - Research Site, Nevers
  - Research Site, Nice
  - Research Site, Nîmes
  - Research Site, Oloron-Sainte-Marie
  - Research Site, Paris
  - Research Site, Perpignan
  - Research Site, Pierre-Bénite
  - Research Site, Pontoise
  - Research Site, Quimper
  - Research Site, Rambouillet
  - Research Site, Reims
  - Research Site, Rennes
  - Research Site, Saint-Aubin-lès-Elbeuf
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Saverne
  - Research Site, Soissons
  - Research Site, Strasbourg
  - Research Site, Thonon-les-Bains
  - Research Site, Toulon
  - Research Site, Toulon Armees
  - Research Site, Toulouse
  - Research Site, Valence
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Verdun
  - Research Site, Vesoul
  - Research Site, Vire
- Germany (10):
  - Research Site, Heidelberg, Baden W�rttemberg
  - Research Site, Ulm, Baden-W�rtemberg
  - Research Site, Löwenstein, Baden-W�rttemberg
  - Research Site, Munchen-Gauting, Bavaria
  - Research Site, Harburg, Hamburg
  - Research Site, Essen, North Rhine-Westphalia
  - Research Site, Hemer, North Rhine-Westphalia
  - Research Site, Leipzig, Saxony
  - Research Site, Halle, Saxony-Anhalt
  - Research Site, Gro�hansdorf, Schleswig-Holstein
- Greece (6):
  - Research Site, Athens, Athens
  - Research Site, Heraklio, Crete
  - Research Site, Ioannina, Ioannina
  - Research Site, Pátrai, Patra
  - Research Site, Piraeus, Piraeus
  - Research Site, Thessaloniki, Thessaloniki
- Italy (23):
  - Research Site, Bologna
  - Research Site, Brindisi
  - Research Site, Carpi
  - Research Site, Cattolica
  - Research Site, Cesena
  - Research Site, Cremona
  - Research Site, Faenza
  - Research Site, Fano
  - Research Site, Legnano
  - Research Site, Lido di Camaiore
  - Research Site, Lugo
  - Research Site, Mantova
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Parma
  - Research Site, Perugia
  - Research Site, Ravenna
  - Research Site, Rimini
  - Research Site, S. Giovanni Rotondo
  - Research Site, Saronno
  - Research Site, Sondrio
  - Research Site, Verona
- Portugal (5):
  - Research Site, Lisbon
  - Research Site, Ponta Delgada
  - Research Site, Porto
  - Research Site, Sta.Ma Feira
  - Research Site, V.N: de Gaia
- Spain (31):
  - Research Site, Madrid, Madrid
  - Research Site, Santa Cruz de Tenerife, Tenerife
  - Research Site, A Coruña
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Cabueñes
  - Research Site, Calella
  - Research Site, Castellon
  - Research Site, Córdoba
  - Research Site, Cuenca
  - Research Site, Elche
  - Research Site, Jaén
  - Research Site, León
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Manacor
  - Research Site, Mataró
  - Research Site, Málaga
  - Research Site, Melilla
  - Research Site, Oviedo
  - Research Site, Palma de Mallorca
  - Research Site, Pamplona
  - Research Site, Puerto Real
  - Research Site, Sagunto
  - Research Site, Salamanca
  - Research Site, Santa Cruz de Tenerife
  - Research Site, Seville
  - Research Site, Tudela
  - Research Site, Valencia
  - Research Site, Xàtiva
  - Research Site, Zaragoza
- Turkey (Türkiye) (6):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Gaziantep
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Konya

REFERENCES:
- [Derived] Vergnenegre A, Carrato A, Thomas M, Jernigan C, Medina J, Cruciani G. Real-world healthcare resource utilization in a European non-small cell lung cancer population: the EPICLIN-Lung study. Curr Med Res Opin. 2014 Mar;30(3):463-70. doi: 10.1185/03007995.2013.860373. Epub 2013 Nov 18. PMID 24188056
- [Derived] Carrato A, Vergnenegre A, Thomas M, McBride K, Medina J, Cruciani G. Clinical management patterns and treatment outcomes in patients with non-small cell lung cancer (NSCLC) across Europe: EPICLIN-Lung study. Curr Med Res Opin. 2014 Mar;30(3):447-61. doi: 10.1185/03007995.2013.860372. Epub 2013 Nov 18. PMID 24168104